CLINICAL TRIAL: NCT04069299
Title: Somatostatin Receptor Expression in Poorly-Differentiated Neuroendocrine Carcinomas of the GI Tract: Analysis Using 68Ga-dotatate PET Scan
Brief Title: Use of 68Ga-dotatate PET Scan in Neuroendocrine Carcinoma of the GI Tract
Status: Active, not recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Other Study IDs: MCC-19943
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Neuroendocrine Carcinoma
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — gallium Ga 68 dotatate; Positron-Emission Tomography; Radionuclide Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving PET scan: Participants with metastatic poorly-differentiated neuroendocrine carcinomas of the GI tract
  Interventions: Drug: 68Ga-DOTATATE; Diagnostic Test: Positron Emission Tomography (PET) Scan

INTERVENTIONS:
Drug: 68Ga-DOTATATE — The NETspot kit is 2 vials, Vial 1 contains 40 mcg dotatate, 5 mcg 1,10phenanthroline; 6mcg gentisic acid and 20 mg mannitol. Vial 2 contains 60 mg formic acid, 56.5 mg sodium hydroxide and water for injection
  Other Names: NETspot
Diagnostic Test: Positron Emission Tomography (PET) Scan — PET scan is an imaging test using radioactive tracers.

SUMMARY:
The purpose of the study is to understand the extent and degree of somatostatin receptor expression in poorly differentiated neuroendocrine carcinomas . This may help to make a determination if a radiolabeled somatostatin analog therapy, also referred to as peptide receptor radiotherapy (PRRT), can be a potential alternative in the future. At this time, radiolabeled somatostatin analogs have not been tested in patients with poorly differentiated neuroendocrine carcinomas, and their efficacy in this disease is not well known Understanding the extent and degree of somatostatin receptor expression is important in order to evaluate the potential of radiolabeled somatostatin analog therapy for treatment of poorly differentiated neuroendocrine carcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female ≥ 18 years old
* Histologically confirmed diagnosis of poorly-differentiated neuroendocrine carcinoma of the gastroenteropancreatic tract or unknown primary
* Evidence of measurable disease per RECIST 1.1 on another imagine modality (CT, MRI or FDGPET) with at least 3 tumors >1cm in largest diameter. CT, MRI or Fluorodeoxyglucose (FDG)-PET must have been performed within 2 months of the study scan. (Of note, participants may sign consent for the study prior to scheduling of said CT, MRI or FDG-PET, but will be considered screen failures if the CT/MRI/FDG-PET does not reveal at least 3 tumors >1cm).

Exclusion Criteria:

* Participants with well-differentiated neuroendocrine tumors
* Participants who have undergone 68Ga-dotatate PET scan in the past
* Pregnant women and/or breastfeeding women. Women of child bearing potential must have a negative pregnancy test prior to scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Moffitt Cancer Center's GI Clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Uniformly Positive 68Ga-dotatate PET | Up to 10 months
  Percentage of participants with uniformly positive 68Ga-dotatate PET (positivity defined as SUV uptake > liver for all tumors at least 1cm in size). Note: Standard Uptake Value (SUV) is used to determine activity in PET imaging.

SECONDARY OUTCOMES:
Percentage of Participants with No Uptake to Very High Uptake on PET | Up to 10 months
  Percentage of Participants with no uptake, heterogeneous uptake (tumors showing substantial differences in Somatostatin receptor [SSTR] uptake), low uptake (max SUV≤ liver), moderate uptake (liver<max SUV ≤2x liver, high uptake (max SUV > 2x liver), very high uptake (max SUV≥ kidney or spleen). Note: Standard Uptake Value (SUV) is used to determine activity in PET imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, MD, Principal Investigator — H Lee Moffitt Cancer & Research Institute
Locations (1):
- H Lee Moffitt Cancer & Research Institute, Tampa, Florida, United States